CLINICAL TRIAL: NCT06805227
Title: Impact of Kinesiology Tape on Quadriceps Muscle: a Randomized Controlled Trial
Brief Title: Effect of Kinesiology Tape on Quadriceps Strength and Performance in Female Futsal Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Norah A. Alshehri, consultant and associate professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: No. KSU-HE-23-091
Record Dates: First submitted 2025-01-22; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Muscle Strength; Rehabilitation; Quadriceps Muscle
Keywords: Kinesiology Tape; Muscle Efficiency; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm: Kinesiology Tape Intervention (Experimental): Description: Participants in this arm received kinesiology tape applied to the dominant leg targeting the rectus femoris, vastus medialis, and vastus lateralis muscles. The tape was applied with a 50% tension level and remained in place for 30 days. Assessments of quadriceps strength and lower limb function were conducted pre- and post-intervention.
  Purpose: To evaluate the effect of kinesiology tape on quadriceps muscle performance.
  Interventions: Other: Kinesiology Tape Application
- Control Arm: No Intervention (No Intervention): Description: Participants in this arm did not receive any kinesiology tape or similar interventions. Their quadriceps strength and lower limb function were assessed at the same intervals as the experimental group for comparison purposes.
  Purpose: To serve as a baseline to compare the effects of the kinesiology tape intervention.

INTERVENTIONS:
Other: Kinesiology Tape Application — Application Area: Applied specifically to the dominant leg, targeting the rectus femoris, vastus medialis, and vastus lateralis muscles.
  Tension Level: Applied with a standardized 50% tension. Duration: The tape was kept in place continuously for 30 days. Color: A blue-colored kinesiology tape was used to standardize the intervention and eliminate potential psychological effects of tape color.
  Technique: Applied by a licensed physical therapist with expertise in kinesiology taping techniques, certified by the Saudi Commission for Health Specialties.
  Arms: Experimental Arm: Kinesiology Tape Intervention

SUMMARY:
The purpose of this randomized controlled trial is to investigate whether kinesiology tape improves quadriceps muscle efficiency in female futsal players. The study aims to answer whether the application of kinesiology tape enhances lower limb function, isometric strength, and eccentric/concentric strength compared to no intervention.

DETAILED DESCRIPTION:
This study explores the potential benefits of kinesiology tape in improving quadriceps muscle performance in female futsal players, a demographic actively engaged in high-intensity sports. The trial was designed to provide robust evidence on whether kinesiology tape can enhance functional and physical performance of the lower limb, addressing a gap in sports medicine research.

The study involved 12 players participating in the Saudi Universities Sports Federation (SUSF) Futsal Championship. Participants were randomly assigned to two groups: an experimental group receiving kinesiology tape intervention and a control group with no intervention. The intervention was conducted over 30 days, with a focus on assessing the impact of kinesiology tape on the dominant leg, targeting key muscles like the rectus femoris, vastus medialis, and vastus lateralis.

To ensure comprehensive evaluation, participants underwent assessments using validated tools for lower limb function, isometric strength, and dynamic strength (eccentric/concentric). These tools included the Single-Leg Hop Test, a hand-held dynamometer, and the Biodex System, which provided precise and reliable measurements of muscle performance.

ELIGIBILITY:
Inclusion Criteria:

* Female futsal players
* Body Mass Index (BMI): 18.5-25 kg/m2.
* Regular participation in sports activities.
* No history of kinesiology tape application on the thighs within six months prior to the study.

Exclusion Criteria:

* Medical history of knee or back pain, lower-limb surgeries, or joint deformities.
* Known allergies to kinesiology tape or conditions such as diabetes, fragile skin, pregnancy, open wounds, or deep vein thrombosis.
* Recent muscular injuries of the lower limbs within six months prior to the study.
* Any other conditions or contraindications that could interfere with participation or the outcomes of the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Effect of Kinesiology Tape on Quadriceps Muscle Strength and Performance in Female Futsal Players | From baseline assessment (pre-intervention) to 30 days post-intervention.
  Isometric Quadriceps Strength: Unit of Measure: Newtons (N). Description: Maximum isometric quadriceps strength of the dominant leg. Assessment Method: Measured using a digital hand-held dynamometer. Participants are seated with their hips flexed at 90° and knees bent at 60°. Maximum force is recorded from three trials of isometric contraction, each lasting five seconds, with a 30-second rest interval between trials.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared due to privacy concerns and the study protocol not including provisions for data sharing.